CLINICAL TRIAL: NCT01069159
Title: Propranolol Treatment of Traumatic Memories (PTTM)
Acronym: PTTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mela, Mansfield, M.D. (Individual)
Responsible Party: Dr. Robin Menzies, Knox Manse
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 505-2010
Record Dates: First submitted 2010-02-13; First posted 2010-02-17 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Traumatic Memory; Posttraumatic Stress Disorder
Keywords: Traumatic memory; Traumatic memories; Traumatic memories and associated symptoms; Posttraumatic Stress Disorder; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol (Active Comparator): The protocol of the study requires that two doses of propranolol (regular propranolol 40 mg followed two hours later by long-acting propranolol 60 mg) be given at the first visit, to be taken within one hour of the reactivation of the traumatic memory. Half of the subjects (33) will be randomized to receive propranolol.
  Interventions: Drug: Propranolol Hydrochloride
- Placebo (Placebo Comparator): The protocol of the study requires that two doses of placebo be given at the first visit, to be taken within one hour of the reactivation of the traumatic memory. Half of the subjects (33) will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol Hydrochloride — The protocol of the study requires that two doses of propranolol (regular propranolol 40 mg followed two hours later by long-acting propranolol 60 mg) or placebo be given at the first visit, to be taken within one hour of the reactivation of the traumatic memory. Subjects will be randomized in a 1:1 ratio to either Propranolol treatment or placebo.
  Other Names: APO-PROPRANOLOL (DIN 00402753); INDERAL LA (DIN 02042231); PROPRANOLOL; PROPRANOLOL LONG-ACTING
  Arms: Propranolol
Drug: Placebo — The protocol of the study requires that two doses of placebo be given at the first visit, to be taken within one hour of the reactivation of the traumatic memory. Half of the subjects (33) will be randomized to receive placebo.
  Arms: Placebo

SUMMARY:
This study will compare the responses of subjects with traumatic memories of varying vintages to either propranolol or placebo in a double-blind setting. It is hypothesized that those subjects who receive propranolol will experience less emotional distress when the memory is subsequently reactivated and less spontaneous re-experiences.

DETAILED DESCRIPTION:
Traumatic memories are responsible for significant emotional distress and disability. They are a cardinal feature of Posttraumatic Stress Disorder (PTSD). Re-experiencing the original traumatic event in a number of different ways (e.g. nightmares, intrusive recollections and dissociative flashbacks) is accompanied by distressing symptoms. The reconsolidation theory of memory proposes that when long-term memories are reactivated, they remain labile for several hours before conversion back to long-term memory. During this period they are susceptible to amnestic agents, like propranolol.

Propranolol Hydrochloride will be compared to placebo in subjects who have emotional distress associated with re-experiences of traumatic events, whether in the context of PTSD or not. Two doses of propranolol or two doses of placebo will be given at the first visit.

The objective of the trial is to determine the effectiveness of brief treatment with propranolol on subjects with traumatic memories and associated symptoms. The research hypothesis is that propranolol will be more effective than placebo, as determined by the measures used, and that this positive outcome will support the reconsolidation theory of memory.

The subjects will undergo clinician rated assessments/scales to determine the presence of pre-treatment mental disorders. Subjects will complete self-rating measures/scales to determine the impact of the traumatic experience. Blood pressure and pulse rates will also be recorded.

Post-treatment outcomes using the same instruments to determine changes at four weeks will be recorded. The differences will be compared and subjected to statistical analysis.

There is an optional component of the study for subjects allocated to the placebo group. At the end of the study, these subjects will be given the opportunity of taking two doses of propranolol and attending a single follow-up session four weeks later for a further interview, rating scale and questionnaire completion. This will provide the subjects who were on placebo an opportunity of possibly benefiting from the active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults between 18 and 70 years of age
* A traumatic memory, as an isolated symptom or in the context of Post-traumatic Stress Disorder

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Current treatment with either a beta-blocker or a corticosteroid medicine
* Medical contraindications, as outlined in the Compendium of Pharmaceutical and Specialties and the Product Monograph
* Subjects who want to retain every aspect of their memory for the traumatic event, as some memory could be lost

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be changes between the pretreatment and posttreatment scores in the Clinician Assessment Posttraumatic Scale (CAPS), Impact of Event Scale (IES) and Traumatic Memory Description Measure (TMDM) instruments. | Visit 2 (Week 4)

SECONDARY OUTCOMES:
The secondary endpoint will be changes between the treatment and posttreatment score in the other scales used - MINI, ZAS, ZDS and NIHS. | Visit 2 (Week 4)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Menzies, MBBS FRCPsych (UK) FRCP (C), Principal Investigator
Locations (1):
- Knox Manse, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Brunet A, Orr SP, Tremblay J, Robertson K, Nader K, Pitman RK. Effect of post-retrieval propranolol on psychophysiologic responding during subsequent script-driven traumatic imagery in post-traumatic stress disorder. J Psychiatr Res. 2008 May;42(6):503-6. doi: 10.1016/j.jpsychires.2007.05.006. Epub 2007 Jun 22. PMID 17588604
- [Background] Nader K, Schafe GE, Le Doux JE. Fear memories require protein synthesis in the amygdala for reconsolidation after retrieval. Nature. 2000 Aug 17;406(6797):722-6. doi: 10.1038/35021052. PMID 10963596
- [Background] Pitman RK. Post-traumatic stress disorder, hormones, and memory. Biol Psychiatry. 1989 Jul;26(3):221-3. doi: 10.1016/0006-3223(89)90033-4. No abstract available. PMID 2545287
- [Background] Pitman RK, Sanders KM, Zusman RM, Healy AR, Cheema F, Lasko NB, Cahill L, Orr SP. Pilot study of secondary prevention of posttraumatic stress disorder with propranolol. Biol Psychiatry. 2002 Jan 15;51(2):189-92. doi: 10.1016/s0006-3223(01)01279-3. PMID 11822998
- [Background] Vaiva G, Ducrocq F, Jezequel K, Averland B, Lestavel P, Brunet A, Marmar CR. Immediate treatment with propranolol decreases posttraumatic stress disorder two months after trauma. Biol Psychiatry. 2003 Nov 1;54(9):947-9. doi: 10.1016/s0006-3223(03)00412-8. PMID 14573324